CLINICAL TRIAL: NCT03055026
Title: Rivaroxaban or Placebo for Extended Antithrombotic Prophylaxis After Laparoscopic Surgery for Colorectal Cancer: a Randomized, Double Blind, Placebo-controlled Study.
Brief Title: Rivaroxaban or Placebo for Extended Antithrombotic Prophylaxis After Laparoscopic Surgery for Colorectal Cancer.
Acronym: PRO-LAPSII
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fadoi Foundation, Italy (Other)
Collaborators: University Of Perugia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FADOI.01.2016
Record Dates: First submitted 2017-02-13; First posted 2017-02-16 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-02

CONDITIONS: Prevention of Venous Thromboembolism
MeSH Terms: interventions — Rivaroxaban

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rivaroxaban (Experimental): Orally administered, at the dose of 10 mg OD for 3 weeks (extended prophylaxis)
  Interventions: Drug: Rivaroxaban
- Placebo (Placebo Comparator): Orally administered, OD for 3 weeks (extended prophylaxis)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rivaroxaban — Tablets
  Arms: Rivaroxaban
Drug: Placebo — Tablets
  Arms: Placebo

SUMMARY:
Rivaroxaban or placebo for extended antithrombotic prophylaxis after laparoscopic surgery for colorectal cancer: a randomized, double blind, placebo-controlled study.

ELIGIBILITY:
Inclusion Criteria:

* Objective diagnosis of colorectal cancer;
* Elective laparoscopic surgery for colorectal cancer
* Whatever the stage of cancer
* Antithrombotic prophylaxis with LMWH administered for 7±2 days after surgery

Exclusion Criteria:

* Age < 18 years
* Surgery for non-cancer disease
* Duration of surgery < 45 min
* Conversion to open surgery
* Other indication for anticoagulant therapy
* Known cerebral metastases
* Kidney or liver failure
* Known hemorrhagic diathesis or high risk for bleeding
* History of intracerebral bleeding or neurosurgery within 6 months
* History of heparin induced thrombocytopenia
* Pregnancy or lactation
* Refusal of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 582 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2021-07-09 (Actual); Study Completion 2021-09-06 (Actual)

PRIMARY OUTCOMES:
Venous thromboembolism | 28±2 days from planned laparoscopic surgery for colorectal cancer in patients randomized to rivaroxaban or placebo.
  The primary study outcome is a composite of symptomatic objectively confirmed VTE, asymptomatic ultrasonography-confirmed DVT or VTE-related death.

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Campanini, Study Director — FADOI Foundation
Locations (17):
- Italy (17):
  - Ospedale Santa Maria delle Grazie, Pozzuoli, Napoli
  - Ospedale di Cittadella, Cittadella, Padova
  - Ospedale San Matteo degli Infermi, Spoleto, Perugia
  - Ospedale E. Agnelli, Pinerolo, Torino
  - Ospedale San Giacomo Apostolo, Castelfranco Veneto, Treviso
  - Istituto Clinico Humanitas Mater Domini, Castellanza, Varese
  - Ospedale San Donato, Arezzo
  - AOU Careggi, Florence
  - Nuovo Ospedale "San Giovanni Battista", Foligno
  - AOU Federico II, Napoli
  - IRCCS Fondazione Pascale, Napoli
  - Policlinico di Padova, Padua
  - Ospedale Santa Maria della Misericordia, Perugia
  - Ospedale San Salvatore, Pesaro
  - Ospedale di Piacenza, Piacenza
  - Policlinico Gemelli, Roma
  - Ospedale Santa Maria, Terni

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Becattini C, Pace U, Pirozzi F, Donini A, Avruscio G, Rondelli F, Boncompagni M, Chiari D, De Prizio M, Visona A, De Luca R, Guerra F, Muratore A, Portale G, Milone M, Castagnoli G, Righini M, Martellucci J, Persiani R, Frasson S, Dentali F, Delrio P, Campanini M, Gussoni G, Vedovati MC, Agnelli G. Rivaroxaban vs placebo for extended antithrombotic prophylaxis after laparoscopic surgery for colorectal cancer. Blood. 2022 Aug 25;140(8):900-908. doi: 10.1182/blood.2022015796. PMID 35580191